CLINICAL TRIAL: NCT00561314
Title: An Evaluation of Focal Ablation Therapy Using High-Intensity Focused Ultrasound in the Treatment of Localized Adenocarcinoma of the Prostate
Brief Title: High-Intensity Focused Ultrasound Ablation in Treating Patients With Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College London Hospitals (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000574344; UCLCTC-UCLH-FOCAL-HIFU; EU-20773
Record Dates: First submitted 2007-11-17; First posted 2007-11-20 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-07

CONDITIONS: Prostate Cancer; Sexual Dysfunction; Urinary Incontinence
Keywords: sexual dysfunction; urinary incontinence; adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Sexual Dysfunction, Physiological; Urinary Incontinence | interventions — Biopsy; High-Intensity Focused Ultrasound Ablation; Magnetic Resonance Spectroscopy

INTERVENTIONS:
Other: questionnaire administration
Procedure: biopsy
Procedure: high-intensity focused ultrasound ablation
Procedure: magnetic resonance imaging
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Highly focused ultrasound energy may be able to kill tumor cells by heating the tumor without affecting the surrounding tissue.

PURPOSE: This phase II trial is studying the side effects and how well highly focused ultrasound energy works in treating patients with localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate feasibility, side effect profile, and patient acceptability of high-intensity focused ultrasound ablation in patients with organ-confined, MRI and histologically proven adenocarcinoma of the prostate.

Secondary

* To determine the effectiveness of therapy via biopsy, MRI, PSA level and estimated time to PSA nadir, and by recording the need for secondary or adjuvant treatment following therapy.

OUTLINE: A probe is inserted into the rectum. High-intensity focused ultrasound (HIFU) energy using the Sonablate system is delivered to the prostate tissue over approximately 2 hours. Patients are then evaluated over a 12-month period.

Patients undergo multi-sequence MRI within 10-20 days after HIFU to assess the extent and volume of tumor necrosis and again at 6 months to assess for disease recurrence. Blood is collected for PSA levels at baseline and then at 1, 3, 6, 9, and 12 months. Patients also undergo transrectal ultrasound biopsy at 6 months to evaluate disease response.

Patients complete questionnaires at baseline and at 1, 3, 6, 9, and 12 months to evaluate erectile and sexual function, urinary flow and continence, and quality-of-life.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Low-risk disease, as defined by the following criteria:

    * Gleason grade total ≤ 7 (patterns 3+4 or 4+3 or less acceptable)
    * Localized disease (unilateral or bilateral) (stage T2c, N0, M0 or less)
    * Serum PSA ≤ 15 ng/mL
* Prostate volume ≤ 40 cc or maximum anterior-posterior length ≤ 40 mm
* Multi-sequence-MRI and transperineal template 5 mm-spaced biopsies performed within the past 6 months
* All malignant areas must be treatable by focal ablation so that approximately 50% of prostate tissue is destroyed and ≥ 1 neurovascular bundle is preserved
* No intraprostatic calcifications making high-intensity focused ultrasound of focal areas of cancer untreatable
* No metastatic disease

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 5 years
* Must be fit for general or regional anesthesia as assessed by Consultant Anesthetist
* No prior rectal fistula
* No American Society of Anesthesiology grades III-IV
* No latex allergies
* No contraindication to MRI scanning (e.g., severe claustrophobia, permanent cardiac pacemaker, or metallic implant likely to contribute significant artifact to images)
* No moderate to severe inflammatory bowel disease

PRIOR CONCURRENT THERAPY:

* No androgen suppression treatment within the past 6 months
* No transurethral resection of the prostate or laser prostatectomy within the past 5 years
* No prior treatment (i.e., radiotherapy, brachytherapy, surgery, laser therapy, chemotherapy, high-intensity focused ultrasound, cryosurgery, thermal therapy, or microwave therapy) for prostate cancer
* No prior significant rectal surgery preventing insertion of transrectal probe

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-02 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Feasibility, patient acceptability and side effect profile of high-intensity focal ultrasound ablation as determined by adverse events
Patient acceptability, urinary symptoms, and erectile function as assessed by Functional Assessment of Cancer Treatment-Prostate (FACT-P); Item International Index of Erectile Dysfunction (IIEF-15); International Prostate Symptom Score (IPSS); I ...

SECONDARY OUTCOMES:
Effectiveness of high-intensity focal ultrasound ablation to control prostate cancer as determined by time to PSA nadir, MRI at 10-20 days and again at 6 months, biopsies of treated areas at 6 months, and by recording the need for secondary or adjuva ...

CONTACTS AND LOCATIONS:
Overall Officials: Mark Emberton, MD, FRCS, MBBS, Study Chair — University College London Hospitals
Locations (2):
- United Kingdom (2):
  - Basingstoke and North Hampshire NHS Foundation Trust, Basingstoke, England
  - University College of London Hospitals, London, England

REFERENCES:
- [Result] Ahmed HU, Hindley RG, Dickinson L, Freeman A, Kirkham AP, Sahu M, Scott R, Allen C, Van der Meulen J, Emberton M. Focal therapy for localised unifocal and multifocal prostate cancer: a prospective development study. Lancet Oncol. 2012 Jun;13(6):622-32. doi: 10.1016/S1470-2045(12)70121-3. Epub 2012 Apr 17. PMID 22512844